CLINICAL TRIAL: NCT06202885
Title: A Comparative Study of Retrospective Outcomes Including Efficacy of Therapy Between Advanced Immunotherapy and Classical Immunochemotherapy in Relapsed/Refractory Lymphoma
Brief Title: CAREMM-2306: Advanced Immunotherapy vs. Classical Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Sung-Soo Park, clinical professor, Seoul St. Mary's Hospital
Other Study IDs: XC23RIDI0102
Record Dates: First submitted 2023-12-18; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T cell engager
  Interventions: Drug: Immunotherapy
- Standard-of-care
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Immunotherapy

SUMMARY:
The goal of this retrospective study is to compare between the case cohort and control cohort.

The case cohort consists of lymphoma patients treated with novel immunotherapy regimen including Chimeric antigen receptor T cell therapy, bispecfic antibody, and/or antibody-drug conjugate.

The control cohort consists of lymphoma patients who received conventional chemotherapy as standard-of-care

The main question[s] it aims to answer are:

* Survival times
* Response outcomes

DETAILED DESCRIPTION:
1. Primary endpoints Comparison of survival time by treatment between two groups
2. Secondary endpoints 2.1 Comparison of progression-free survival between two groups 2.2 Comparison of response rates between two groups 2.3 Comparison of input medical costs between two groups.

2. Study subjects: Patients treated for lymphoma at Yeouido St. Mary's Hospital and Seoul St. Mary's Hospital (Both are located on Seoul, Korea) between May 2009 and June 2023.

3. Selection criteria: 3.1 Patients diagnosed with malignant lymphoma at Catholic Yeouido St. Mary's Hospital and Seoul St. Mary's Hospital between May 2009 and June 2023.

3.2 Age 19 or older. 3.3 Patients who treated with salvage chemotherapy for the relapsed/refractory lymphoma.

4. Exclusion criteria: 4.1 Patients suffering from acute leukemia. 4.2 Patients additionally diagnosed with solid cancer (colon cancer, lung cancer, stomach cancer, etc.) during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with malignant lymphoma at Catholic Yeouido St. Mary's Hospital and Seoul St. Mary's Hospital between May 2009 and June 2023.
2. Age 19 or older.
3. Anti-cancer salvage chemotherpay for the treatment of relapsed/refractory lymphoma.

Exclusion Criteria:

1. Patients suffering from acute leukemia.
2. Patients additionally diagnosed with solid cancer (colon cancer, lung cancer, stomach cancer, etc.) during treatment.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated for lymphoma at Catholic Yeouido St. Mary's Hospital and Seoul St. Mary's Hospital from May 2009 to June 2023
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Survival Periods Among Groups Comparison of Survival Periods Among Groups | Time Frame: Up to 2 years
  overall survival

SECONDARY OUTCOMES:
Comparison of Progression-Free Survival Periods | Time Frame: Up to 2 years
  progression-free survival

OTHER OUTCOMES:
Comparison of Response Rates | Time Frame: Up to 2 years
  response rate
Comparison of Healthcare Costs | Time Frame: Up to 2 years
  costs

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No